CLINICAL TRIAL: NCT02718183
Title: Effect on Periodontal Markers Interleukin-RANK by Walking Bleaching Non-Vital Technique: Clinical Randomized Double-blind Trial
Brief Title: Effect on Periodontal Markers by Bleaching Intracoronal Technique
Acronym: BLEIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 03/16
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Discolored Teeth
MeSH Terms: conditions — Tooth Discoloration | interventions — Hydrogen Peroxide; Carbamide Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PH (Experimental): Hydrogen peroxide 35% to intracoronal bleaching in discoloration teeth eith endodontic treatment
  Interventions: Other: Hydrogen Peroxide 35% (Opalescence Endo - Ultradent, USA)
- PC (Experimental): Carbamide peroxide 37% to intracoronal bleaching in discoloration teeth eith endodontic treatment
  Interventions: Other: carbamide peroxide 37% (Whiteness Superendo, FGM, Brazil).

INTERVENTIONS:
Other: Hydrogen Peroxide 35% (Opalescence Endo - Ultradent, USA) — bleaching teeth gel to intracameral use.
  Other Names: Hp 35%
  Arms: PH
Other: carbamide peroxide 37% (Whiteness Superendo, FGM, Brazil). — bleaching teeth gel to intracameral use.
  Other Names: Cp 37%
  Arms: PC

SUMMARY:
OBJECTIVES: The aim of this clinical randomized, double-blind clinical study was to assess the markers levels of RANKL IL-1B and OPGL, involved in the external cervical resorption as a primary outcome, and change color effectiveness in patients undergoing intracoronary bleaching.

METHOD: 46 volunteers (50 teeth) participated with discoloration on non-vital teeth, with the endodontic treatment in good condition. Patients were randomly located into two study groups according to product G1 = 35% hydrogen peroxide (n = 25) and G2 = 37% carbamide peroxide (n = 25).

The intracameral bleaching was performed with a walking bleaching technique of 4 sessions Gingivocrevicular transudate samples were taken to determine levels of Il1b, RANKL, and OPGL with absorbent paper (Periopaper®), they are obtained from six sites per tooth bleaching: 3 vestibular and three palatine (mesial, middle and distal), in 6 opportunities:

Baseline, after 4-sessions of intracameral bleaching and a one week after treatment. Total proteins are quantified by Bradford ® system and from the eluted sample of RANKL, IL 1b and OPGL levels measured by ELISA (Quantikine®; R&D Systems Inc.).

The color was evaluated in each session with Vita EasyShade spectrophotometer is used with the CIEL*a*b system to measure the total variation in color (ΔE), between the baseline and the different evaluation times.

DETAILED DESCRIPTION:
The trial was randomized and double-blind (patient and operator). Advertising was held to invite participation in dental school and through social networks like Facebook or Twitter.

Sample size

To determine the size of the sample GPower 3.1 software was used, considering a significance level of 5% statistical power of 80%.

A total of 74 patients were examined to assess whether they met the criteria for inclusion and exclusion. Patients: over 18 years, with one or more non-vital teeth, the restoration does not cover the vestibular face, endodontic treatment is in good condition, without apical lesion, with no previous experience of tooth whitening and tooth shade A2 or greater according to the Vita Classical scale. Patients were excluded pregnant or lactating, patients with enamel hypoplasia, with teeth stained by tetracycline or fluorosis, in orthodontic treatment with fixed appliances, patients with cancer or periodontal diseases. In addition to those volunteers to be examined clinically and radiographically present caries, periapical lesions, external or internal dental resorption and / or periodontal disease, as may be informed and referred to specialists for treatment.

46 patients, of whom 44 completed treatment and attended all controls were selected.

Were formed at randomization two study groups as the bleaching agent used, each with teeth n = 25, G1 = teeth bleached with Hydrogen Peroxide 35% (Opalescence Endo - Ultradent, USA). G2 = bleached teeth with carbamide peroxide 37% (Whiteness Superendo, FGM, Brazil).

Bleaching procedure

The application of the bleaching agents was performed according to manufacturers instructions in four sessions with an outpatient technique (Walking Bleaching), with one week apart from each.

Session Preparation: Preparing root canal with absolute isolation, were removed from 3mm seal the endodontic cement-enamel limit reference. The final sealing was made with 2mm with glass ionomer resin composite modificao and curing by (Riva Light Cure, SDI, Australia) and light-cured for 40 seconds (Cal Radii, SDI, Australia).

Unblocking a radiographic control and sealing the root canal, and radiographs, post seal was obtained.

4 sessions of Whitening: The Application of the bleaching agent was according to manufacturer's instructions. An amount of gel bleaching agent was left intracamerally with moisture (Walking Bleaching). Subsequently he sealed with a temporary cement to the next session.

Closing session: the access cavity was washed with water and a temporary sealing leave for 7 days prior to the completion of the final seal.

Patients were advised not to eat or drink foods that can stain, such as coffee, tea, red wine, etc. during the study period. They were given written instructions and contact information for any questions or problems arise.

Color Evaluation

Two calibrated evaluators, with 80% agreement (Kappa test), recorded the color of teeth at baseline (baseline), immediately after each bleaching session, one week and one month post-treatment.

Color evaluation was measured in the middle third of the labial surface of tooth bleaching. Patients were examined in the same room with the same lighting, for both examiners independently. using the Vita Bleachguide scale (Vita Zahnfabrik, Bad Säckingen, Germany) .For every "value" color is assigned a numerical value in order to calculate the change in units scale (SGU Δ).

Evaluation of markers RANKL-OPG-Interleukin in crevicular gingival fluid (FGC) Obtaining and handling of samples FGC

FGC samples were obtained from six sites periodontal 3 vestibular and 3 palatal / lingual (average mesial - distal) undergoing teeth whitening. Samples were taken before the whitening (baseline) and after each whitening session, a week and a month post-whitening.

For this were used Periopaper® absorbent paper strips (OraFlow Inc., New York, NY, USA). The teeth were isolated from a relative fashion using cotton rolls, once isolated with a Gracey 3/4 the supra-gingival plaque be removed and gently the surface of the triple air dry syringe. The paper strip was introduced into the selected tooth gingival sulcus until mild resistance tissue and held for 30 seconds. Then they were placed in properly labeled Eppendorf tubes and transported immediately to be stored at -80 ° C until the centrifugal elution process. The paper strips contaminated with saliva or blood were discarded.

The paper strips were subjected to centrifugal elution to obtain total proteins present in the FGC. To do this, incubated for 30 minutes in 100 .mu.l of elution buffer containing 0.05% Tween in Tris-HCl pH 7.4 (Fluka, Sigma-Aldrich Chemie GmbH, Buchs, Switzerland) and then centrifugarnn 10,000 xg for 5 minutes at 4 ° C. The process of centrifugal circumvention repetio 3 times to a final volume of 300 ul, which was stored at -80 ° C until analysis.

Evaluation of markers RANKL-OPG-Interleukin in crevicular gingival fluid (FGC) Total proteins were quantified by the Bradford ® system (R & D Systems Inc., Minneapolis, MN, USA) and from 50 ul of sample eluted from medieronn levels of RANKL, OPG and interleukin by ELISA (Quantikine®; R & D Systems Inc. ) following the manufacturer's protocol. The average absorbance at 492 nm with correction at 630 nm using an automated plate reader (Universal ELx800 Microplate Reader, Bio-Tek Instruments Inc., Winooski, VT, USA). The concentration of the markers in each sample was calculated using an equation of the line of 4th grade.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* with one or more non-vital teeth,
* the restoration does not cover the vestibular face of teeth,
* endodontic treatment is in good condition, without apical lesion,
* with no previous experience of tooth whitening and tooth shade A2 or greater according to the Vita Classical scale.

Exclusion Criteria:

* excluded pregnant or lactating,
* patients with enamel hypoplasia,
* with teeth stained by tetracycline or fluorosis,
* in orthodontic treatment with fixed appliances,
* patients with cancer or periodontal diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Bone destruction markers in gingival fluids | 1 year
  [Interleukin 1b , RANK-L, OPG ] (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: eduardo fernandez, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miranda CB, Mayer C, Ledezma P, Vernal R, Rivera O, Godoy EF. Persistent Inflammatory Response in Periodontal Tissues After Walking Bleach: A Clinical Biomarker-Based Study. Aust Endod J. 2025 Dec;51(3):619-631. doi: 10.1111/aej.12975. Epub 2025 Jul 16. PMID 40667613
- [Derived] Bersezio C, Martin J, Mayer C, Rivera O, Estay J, Vernal R, Haidar ZS, Angel P, Oliveira OB Jr, Fernandez E. Quality of life and stability of tooth color change at three months after dental bleaching. Qual Life Res. 2018 Dec;27(12):3199-3207. doi: 10.1007/s11136-018-1972-7. Epub 2018 Aug 21. PMID 30132252